CLINICAL TRIAL: NCT03641677
Title: Increasing Lung Transplant Availability Using Normothermic Ex Vivo Lung Perfusion (EVLP) at a Dedicated EVLP Facility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lung Bioengineering Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EVP-DEV-LTX-301
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Lung Diseases
Keywords: EVLP; ex vivo lung perfusion; organ perfusion; CLES; centralized lung evaluation system; united therapeutics
MeSH Terms: conditions — Lung Diseases | interventions — Lung Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- EVLP (Experimental)
  Interventions: Device: Centralized Lung Evaluation System; Procedure: Lung Transplant
- Control (Active Comparator)
  Interventions: Procedure: Lung Transplant

INTERVENTIONS:
Device: Centralized Lung Evaluation System — Assessment of allograft lung for transplant suitability
  Arms: EVLP
Procedure: Lung Transplant — Orthotopic single or double lung transplantation.

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the Centralized Lung Evaluation System (CLES) in enabling evaluation of potential donor lungs not otherwise used for transplant into subjects with end stage, survival-limiting lung disease in need of lung transplantation. This will be accomplished by evaluating subject survival at the later of 12 months or hospital discharge post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* Aged 18 years or older;
* Informed consent is given for participation in the Study by the patient or patient's designated representative; and
* Patient undergoes lung transplantation.

Exclusion Criteria:

* Patients listed for same-side lung re-transplantation.
* Patients listed for multiple organ transplantation including lung and any other organ.
* Patients listed for live donor lobar lung transplant.
* Patients positive for human immunodeficiency virus (HIV) or Burkholderia cenocepacia infection.
* Patient receives a standard of care (non-EVLP) lung transplant but does not match to an EVLP subject based on the criteria for control matching.
* Participating in another interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
12 month survival | 12 months

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Mayo Clinic Florida, Jacksonville, Florida
  - Emory University Hospital, Atlanta, Georgia
  - University of Maryland Medical System, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - NYU Langone Health, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - INOVA Fairfax Hospital, Falls Church, Virginia